CLINICAL TRIAL: NCT04423614
Title: Telehealth-Delivered Preoperative Inspiratory Muscle Training: An Innovative Solution to Conserve Scarce ICU Resources
Brief Title: Preoperative Inspiratory Muscle Training
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study staff were busy with other projects and unable to devote time to this study
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB202001038; OCR35362 (Other: UF OnCore)
Record Dates: First submitted 2020-06-02; First posted 2020-06-09 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Mechanical Ventilation Complication
Keywords: Mechanical ventilation; Inspiratory muscle training; Difficulty weaning from mechanical ventilation

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into one of two arms. In Arm 1, subjects will perform pre-operative inspiratory muscle training. In Arm 2, subjects will perform pre-operative relaxation breathing. A diaphragm biopsy will be taken during surgery for both arms and the tissue will be compared. In addition, a biopsy of the pectoralis major will be obtained from each subject and serve as a non-exercised control which will compared to the subject's diaphragm muscle biopsy (which participated in the intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training (IMT) (Experimental): Pre-operative inspiratory muscle training
  Interventions: Other: Inspiratory Muscle Training
- Relaxation Breathing (RLX) (Experimental): Relaxation breathing exercises
  Interventions: Other: Relaxation Breathing

INTERVENTIONS:
Other: Inspiratory Muscle Training — Inspiratory muscle training exercises, performed 5 times a week for 2-4 weeks prior to cardiac surgery.
  Arms: Inspiratory Muscle Training (IMT)
Other: Relaxation Breathing — Relaxation breathing exercises, performed 5 times a week for 2-4 weeks prior to cardiac surgery.
  Arms: Relaxation Breathing (RLX)

SUMMARY:
In light of the corona virus pandemic (COVID-19), there is critical need to conserve scarce mechanical ventilation (MV) resources. This study evaluates an intervention in non-infected cardiac patients as a means to assist with minimizing MV and ICU length of stay (LOS). Pre-op inspiratory muscle training (IMT) has been shown to decrease pulmonary complications, MV dependence, and ICU LOS following thoracic surgery. The investigators aim to determine the mechanism of remodeling in diaphragms of adults who undergo pre-op IMT.

DETAILED DESCRIPTION:
Highly active muscles such as the diaphragm are particularly sensitive to both disuse and training. For example, diaphragm fibers of controlled mechanically ventilated young adults atrophy by more than 50% within 36 hours of complete inactivity, and mechanical ventilation (MV) initiates signaling pathways within the first several hours of inactivity that promote progressive diaphragmatic fiber dysfunction. The investigators have shown that widespread atrophy signaling begins in the operating room during cardiac surgery, after only a few hours of MV. In addition to this fiber atrophy, MV leads to significant declines in the strength of the diaphragm, which can lengthen the time it takes to wean from MV. The clinical occurrence of early onset, progressive contractile dysfunction is defined as ventilator-induced diaphragmatic dysfunction (VIDD). VIDD is regarded as a primary contributor to difficulties with weaning from MV.

Conversely, the investigators have shown that IMT increases the pressure-generating capacity of the diaphragm and inspiratory synergist muscles, and facilitates weaning in patients with VIDD. Preoperative IMT for as little as 1-2 weeks reportedly increases inspiratory muscle strength. IMT prior to cardiothoracic surgery has been shown to reduce post-operative pulmonary complications such as atelectasis, pneumonia, or delayed ventilator weaning. Additionally, strength gains associated with preoperative IMT are associated with shorter ICU and hospital lengths of stay, which may potentially offer a cost benefit.

Unfortunately, very little is understood about the neuromuscular adaptations and signaling mechanisms that contribute to these IMT clinical advantages. A particularly novel aspect of this project is it will be the first study of the mechanisms that contribute to diaphragm strengthening. A greater understanding of these mechanisms may help future investigators to develop more efficient exercise prescriptions to offset MV use in cases such as surgery, and it may help identify molecules and exercise that could protect the diaphragms of individuals who cannot exercise in advance, as in the case of acute infections that compromise breathing.

The overall objective of this study is to investigate diaphragm neuromuscular remodeling associated with pre-operative, telehealth delivered IMT, compared with relaxation breathing training (RLX). Guided RLX exercises have been shown to improve post-operative pain perception and modestly lower systolic blood pressure in hypertensives but are not thought to significantly alter diaphragm strength.

Forty adult volunteers will receive either IMT (n=20) or RLX training (n=20) for 2-4 weeks prior to elective cardiothoracic surgery and undergo breathing performance tests before and after the training period. A full thickness biopsy (approximately 6mm x 20 mm) from the right ventral costal diaphragm will be acquired as soon as the diaphragm is exposed during surgery. Additionally, a biopsy from the pectoralis major will be obtained and used as a non-exercised control muscle. Histological and RNA sequencing analyses will be performed to examine the mechanisms that contribute to neuromuscular adaptations to training.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery candidate
* Ability to complete pre-operative breathing exercises

Exclusion Criteria:

* Surgery is scheduled in less than 2 weeks
* New York Heart Association Class III or IV Cardiac Disease
* History of hemiparesis
* History of spinal cord injury
* History of progressive neuromuscular disease that may interfere with the ability to complete study interventions
* Previous cardiothoracic surgery within the last 12 weeks
* History of pneumonectomy
* History of lung surgery
* History of skeletal pathology (e.g. scoliosis) that may interfere with chest wall movements
* Routine usage of muscle relaxants, immunosuppressants, or corticosteroid medications within the past 30 days
* Forced expiratory volume 1 less than 40% of age-predicted value
* Presence of active malignancy
* Presence of any organ dysfunction that may limit ability to participate in seated respiratory exercises

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory pressure | Post breathing exercise sessions (up to 4 weeks)
  Maximal inspiratory pressure will be quantified in cm of water pressure.
Muscle fiber cross-sectional area and fiber type proportion. | Intra-operatively
  Histology will be used to determine fiber type and cross-sectional area using primary antibodies for laminin and type-specific myosin heavy chain, followed by a triple immunofluorescence-conjugated secondary antibody labeling technique.

SECONDARY OUTCOMES:
Peak expiratory flow | Post breathing exercise sessions (up to 4 weeks)
  Spirometry will be used to measure peak expiratory flow during a voluntary cough maneuver. It will be quantified in liters per second.
Time to extubation | Up to discharge from ICU
  Time to extubation will be measured as hours of post-operative mechanical ventilation.
Length of ICU stay | Up to 1 month
  Length of ICU stay will be measured as hours spent in ICU after surgery.
Length of hospital stay | Up to 1 month
  Length of hospital stay will be measured as hours spent in hospital after surgery.
Neuromuscular junction morphology | Intra-operatively
  Histology will be used to assess neuromuscular junction number and morphology using immunofluorescent-labeled antibodies for synaptophysin and alpha bungarotoxin. Neuromuscular junction image stacks will be visualized with confocal microscopy and morphology classified according to endplate area and area fractions of fragmented junctions, acetylcholine receptor-occupied endplate area, synaptophysin-occupied endplates, and abandoned endplates.
Muscle differential gene expression | Intra-operatively
  RNA isolation will be performed using Tri Reagent and chloroform based manual method. RNA will be quantified and RNA-Seq will be used to assess gene expression.
Physical Function | Post breathing exercise sessions (up to 4 weeks)
  Physical function will be assessed with the Patient Reported Outcomes Measurement Information System Physical Function questionnaire. Each answer corresponds to a number between 1 and 5.
Dyspnoea | Post breathing exercise sessions (up to 4 weeks)
  Dyspnoea will be assessed with the Dyspnoea 12 Questionnaire. Responses range from None to Severe.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Smith, PhD, PT, Principal Investigator — University of Florida; Thomas Beaver, MD, MPH, Principal Investigator — University of Florida